CLINICAL TRIAL: NCT06707142
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose and Multiple Ascending Dose Trial in Healthy Adult Participants to Evaluate the Safety, Tolerability, and Pharmacokinetics of TBD11 With an Open Label (Single Dose) Food Effect Panel
Brief Title: A Trial in Healthy Adult Participants to Evaluate the Safety, Tolerability, and Behavior in the Body of TBD11
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Gates MRI-TBD11-101
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Healthy Adult Participants
Keywords: Single Ascending Dose; Multiple Ascending Dose; TBD11; Food Effect; Safety; Tolerability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1 Cohort 6 and Part 2, Cohort 4 are Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TBD11 (Experimental): In Part 1 double-blind phase of the trial (SAD), cohorts 1 to 5 and cohort 7 will receive doses of TBD11; 8 participants in each cohort will be randomized (6:2) to receive TBD11 or placebo.
  The FE component of Part 1 (cohort 6) is open-label and 12 participants will receive TBD11 to evaluate the food effect.
  In Part 2, double blind phase of the trial, MAD, 48 participants will be randomized (3:1) to receive TBD11 or placebo in Cohorts 1-3.
  In Part 2 (Cohort 4), all participants will receive open-label TBD11
  Interventions: Drug: TBD11; Drug: Placebo
- Placebo (Placebo Comparator): Participants in Part 1 (cohorts 1-5 and cohort 7) and Part 2 will receive placebos matched to TBD11
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TBD11 — TBD11 will be administered orally.
  Arms: TBD11
Drug: Placebo — Placebo will be administered orally.

SUMMARY:
This is a randomized, double-blind, placebo controlled First in human (FIH) trial of TBD11, administered to healthy adults. The trial will be conducted in two parts. Part 1 will consist of single ascending dose (SAD) and Food effect (FE) cohorts, and Part 2 will consist of multiple ascending dose (MAD) cohorts and tablet formulation evaluation (Part 2, Cohort 4).

ELIGIBILITY:
Inclusion Criteria:

* Is healthy as determined by the Investigator via medical history and clinical examination before enrollment in the trial.
* Can understand and comply with the trial and site procedures, understand the risks involved in the trial, and provide written informed consent before the first trial-specific procedure.
* Can complete all Screening period evaluations and stay in the clinical research facility for the duration of the inpatient periods of the trial.
* Has Body Mass Index (BMI) between 18 and 32 kilograms per meter square (kg/m2), inclusive, and body weight not less than 50 kg at Screening.
* Has resting vital signs within the following ranges at Screening and Day -1:

  1. Systolic blood pressure (SBP) >= 100 millimeters of Mercury (mmHg) and <= 140 mmHg
  2. Diastolic blood pressure (DBP) >= 60 mmHg and <= 90 mmHg
  3. Heart rate between 50 and 100 beats per minute (bpm)
* If individual's assigned sex at birth is female, they must have negative urine and serum pregnancy tests at Screening, and be of non-childbearing potential based on either of the following:

  1. Is post-menopausal defined as amenorrhea for at least 12 months in absence of any exogenous hormonal treatments and follicle stimulating hormone (FSH) levels in the laboratory-defined postmenopausal range, or,
  2. Reports being surgically sterilized (ie, tubal ligation, hysterectomy, bilateral oophorectomy/salpingectomy), and provides written documentation [(ie, medical record(s)], where feasible, to document such procedure(s) to the Principal Investigator. The site must make documented attempts to obtain medical records. If records cannot be retrieved, a participant may be enrolled at the Principal Investigator's discretion.

Exclusion Criteria:

* Has current or past history of a clinically significant cardiovascular, cerebrovascular, respiratory, gastrointestinal, hematologic, renal, hepatic, immunologic, metabolic, urologic, neurologic, dermatologic, psychiatric, or other major disease, as determined by the Investigator.
* Has history of or has clinically relevant cardiovascular disorder, such as heart failure, coronary artery disease, controlled or uncontrolled hypertension, arrhythmia, tachyarrhythmia, prolonged QT syndrome, or presence of symptom(s) strongly suggestive of such a problem, such as exertional chest pressure/pain or unexplained syncope.
* Had an active malignancy within 5 years from Screening, except basal cell or squamous cell skin cancers. Any history of breast cancer or melanoma will be exclusionary.
* Has history of any drug abuse within 1 year prior to Screening or has used any hard drugs (such as cocaine, phencyclidine [PCP], natural and synthetic opiates, and amphetamine derivatives) within 1 year prior to Screening. Individuals that have taken an opioid or amphetamine medication within the previous year prior to Screening that was prescribed by a healthcare provider will not be excluded unless they are currently taking the medication at the time of Screening.
* Had any surgical or medical condition or history that, in the opinion of the Investigator, may potentially alter the absorption, metabolism, or excretion of study treatment, such as, but not limited to, gastric bypass, sleeve, banding surgery, or gastric or duodenal ulcers.

Additional inclusion/exclusion criteria are defined in the protocol.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) after administration of single doses or multiple doses in healthy adult participants | Part (Pt.) 1 (Cohorts 1-5, 7):Day 1-7; Pt. 1 (Cohort 6, Periods [Pds.] 1-3):Day 1 through the washout of each respective Pd.; Pt. 2 (Cohorts 1-3):Day 1-19; Pt. 2 (Cohort 4): Pd.1: Day 1 through last day of washout; Pd.2: Day 1 through last day of washout
Number of participants with clinically significant changes from Baseline in clinical laboratory values | Part (Pt.) 1 (Cohorts 1-5, 7):Day 1-7; Pt. 1 (Cohort 6, Periods [Pds.] 1-3):Day 1 through the washout of each respective Pd.; Pt. 2 (Cohorts 1-3):Day 1-19; Pt. 2 (Cohort 4): Pd.1: Day 1 through last day of washout; Pd.2: Day 1 through last day of washout
  Blood samples will be collected for the analysis of clinical laboratory measures including clinical chemistry, hematology, coagulation, and urinalysis.
Number of participants with clinically significant changes from Baseline in vital signs | Part (Pt.) 1 (Cohorts 1-5, 7):Day 1-7; Pt. 1 (Cohort 6, Periods [Pds.] 1-3):Day 1 through the washout of each respective Pd.; Pt. 2 (Cohorts 1-3):Day 1-19; Pt. 2 (Cohort 4): Pd.1: Day 1 through last day of washout; Pd.2: Day 1 through last day of washout
Number of participants with clinically significant changes from Baseline in Electrocardiogram (ECG) parameters | Part (Pt.) 1 (Cohorts 1-5, 7):Day 1-7; Pt. 1 (Cohort 6, Periods [Pds.] 1-3):Day 1 through the washout of each respective Pd.; Pt. 2 (Cohorts 1-3):Day 1-19; Pt. 2 (Cohort 4): Pd.1: Day 1 through last day of washout; Pd.2: Day 1 through last day of washout
  ECG parameters include heart rate, RR interval, PR interval, QRS duration, QT interval, and QT interval corrected by Fridericia's formula [QTcF].

SECONDARY OUTCOMES:
Part 1: Maximum plasma drug concentration (Cmax) of TBD11 in treated participants | Day 1
  Blood samples are collected at indicated time points for pharmacokinetic (PK) analysis of TBD11. PK parameters are analyzed using standard non-compartmental analysis.
Part 1: Area under the concentration-time curve calculated to last quantifiable observed sample (AUClast) of TBD11 in treated participants | Day 1 through Day 7
Part 1: Terminal elimination half-life (t1/2) of TBD11 in treated participants | Day 1 through Day 7
Part 1: Time to maximal concentration (Tmax) of TBD11 in treated participants | Day 1
Part 2: Cmax of TBD11 in treated participants | Day 1 and Day 14
Part 2: Tmax of TBD11 in treated participants | Day 1 and Day 14
Part 2: Area Under the concentration time curve from Zero to 24 hours (AUC 0-24) of TBD11 in treated participants | Day 1
Part 2: AUC last of TBD11 in treated participants | Day 1 and Day 14
Part 2: Minimum plasma drug concentration (Cmin) of TBD11 in treated participants | Day 14
Part 2: Accumulation ratio (area under plasma concentration-time curve over dosing interval [AUCtau] / AUC0-24) of TBD11 in treated participants | Day 14
Part 2, Cohort 4: Geometric mean ratio (GMR) Cmax,capsules / Cmax,tablets in treated participants | Day 1 through last day of washout of the treatment period
Part 2: Cohort 4: GMR AUC (0-infinity) capsules / AUC(0-inf) tablets | Day 1 through last day of washout of the treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: This will be done within 12 months of the study completion date Access Criteria: Anonymized participant level data may be shared with external researchers in accordance with the trial participants' written and executed informed consent document and any local or applicable regulations on data sharing. Qualified researchers may submit a request for anonymized participant level data along with a research proposal to Gates MRI for review. The types of supporting information that could be shared with external researchers include: the Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report, and analytic code. A data sharing agreement must be in place before any clinical trial data are shared. There are additional circumstances that may prevent the sharing of data with external researchers, including but not limited to contractual obligations to existing partners and any restrictions imposed by regulatory bodies.